CLINICAL TRIAL: NCT00445913
Title: Autologous Dendritic Cell Therapy for Type 1 Diabetes Suppression: A Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0509115; NIDDK R33 DK683044 (Other: NIH NIDDK)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; dendritic cells; cell vaccine; safety; reversal
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control dendritic cells (Experimental): autologous dendritic cells that are not treated
  Interventions: Biological: control dendritic cells
- AS ODN dendrtitic cells (Experimental): autologous dendritic cells treated ex vivo with the mixture of the antisense oligonucleotides
  Interventions: Biological: Diabetes-suppressive dendritic cell vaccine

INTERVENTIONS:
Biological: Diabetes-suppressive dendritic cell vaccine — The dendritic cells will be treated ex vivo with the antisense oligonucleotides and cryopreserved in aliquots for subsequent intradermal administration into sites closest to the physical location of the pancreas inside the body. Physiologic, biologic and immunologic responses to the dendritic cell vaccine will be evaluated over the period of the trial. The first group of volunteers will receive autologous dendritic cells without any ex vivo treatment (7/15) and the second group will be administered iDC (8/15). If there is no evidence of toxicity or adverse events associated with the dendritic cell vaccine, and only upon FDA and IRB approval we will initiate a new study comparing efficacy of control DC and iDC in improving glycemia and reversing autoimmunity in new-onset patients.
  Other Names: diabetes-suppressive dendritic cells
  Arms: AS ODN dendrtitic cells
Biological: control dendritic cells — The dendritic cells will be treated ex vivo with vehicle and cryopreserved in aliquots for subsequent intradermal administration into sites closest to the physical location of the pancreas inside the body. Physiologic, biologic and immunologic responses to these control dendritic cells will be evaluated over the period of the trial. The first group of volunteers will receive autologous dendritic cells without any ex vivo treatment (7/15) and the second group will be administered iDC (8/15). If there is no evidence of toxicity or adverse events associated with the dendritic cell vaccine, and only upon FDA and IRB approval we will initiate a new study comparing efficacy of control DC and iDC in improving glycemia and reversing autoimmunity in new-onset patients.
  Arms: control dendritic cells

SUMMARY:
The proposed studies describe a randomized trial to evaluate the safety of a new diabetes-suppressive cell vaccine, consisting of autologous monocyte-derived dendritic cells treated ex vivo with antisense phosphorothioate-modified oligonucleotides targeting the primary transcripts of the CD40, CD80 and CD86 co-stimulatory molecules (immunoregulatory DC; iDC). The hypothesis to be tested in this study is that iDC are safe and without toxicity in established type 1 diabetic patients.

Fifteen (15) individuals exhibiting fully-established, insulin-dependent type 1 diabetics, without any diabetes-related complications, infectious disease, or other medical anomaly, will be enrolled to establish safety of the approach. 7/15 volunteers will be administered autologous control dendritic cells and 8/15 will be administered iDC. The study is anticipated to be complete by twelve (12) months.

Currently, other than a humanized anti-CD3 antibody with considerable side effects, there is no other means to reverse new-onset type 1 diabetes. These studies will be the first ever to employ autologous dendritic cell transfer to suppress an autoimmune disease and to perhaps reverse it early on in the clinical process.

DETAILED DESCRIPTION:
In this study, volunteers with established type 1 diabetes that requires insulin replacement who do not exhibit any diabetes-related complications or any other clinical pathology will first undergo complete physical, biochemical and immunological evaluation. Monocyte-derived autologous dendritic cells will be obtained following leukapheresis. The dendritic cells will be treated ex vivo with the antisense oligonucleotides and cryopreserved in aliquots for subsequent intradermal administration into sites closest to the physical location of the pancreas inside the body. Physiologic, biologic and immunologic responses to the dendritic cell vaccine will be evaluated over the period of the trial. The first group of volunteers will receive autologous dendritic cells without any ex vivo treatment (7/15) and the second group will be administered iDC (8/15). If there is no evidence of toxicity or adverse events associated with the dendritic cell vaccine, and only upon FDA and IRB approval we will initiate a new study comparing efficacy of control DC and iDC in improving glycemia and reversing autoimmunity in new-onset patients.

Currently, other than a humanized anti-CD3 antibody with considerable side effects, there is no other means to reverse new-onset type 1 diabetes. These studies will be the first ever to employ autologous dendritic cell transfer to suppress an autoimmune disease and to possibly reverse it early on in the clinical process.

We propose to ascertain the safety of autologous dendritic cells treated ex vivo with antisense oligonucleotides targeting the primary transcripts of the CD40, CD80 and CD86 co-stimulatory molecules (we term these cells "immunoregulatory dendritic cells; iDC) first in volunteers with established type 1 diabetes.

Personality traits and emotional stability have been linked to treatment adherence in other medical populations (e.g. Christensen et al, 2002; Dew et al., 2001). In that adherence to this protocol (e.g. remaining in the study) by this small sample will impact significantly on results and that the treatment itself may affect mood, we will assess personality traits at baseline and monitor mood throughout the study period.

2.2 Significance of the studies: We do not anticipate any safety issues with this approach but we must be cautious at all levels given that this is immunomodulation therapy. At the very least, data will be obtained on whether the success we have observed with the iDC in NOD mice can be eventually adapted in other protocols aimed to restore normoglycemia or improve glycemic control along with increased prevalence of putative immunoregulatory T cells in recently-diagnosed humans.

3.0 RESEARCH DESIGN AND METHODS

3.1 Drug/Device Information 3.1.1 Autologous Dendritic Cells (Control Dendritic Cells): These are cells derived from the leukapheresis product of each patient. The leukapheresis product is processed inside an Elutra/AastromTM cell elutriation system (Refer to appended SOP # CPL-0158 and CPL-0166) to obtain immature dendritic cells. The final autologous product after these procedures is termed Control Dendritic Cells.

3.1.2 Autologous Immunoregulatory, Diabetes-Suppressive Dendritic Cells (iDC): We have submitted an IND application (appended) to the FDA to cover a diabetes-suppressive embodiment of Control Dendritic Cells, which we term "immunoregulatory dendritic cells; iDC. The IND covers the treatment of Control Dendritic Cells with phosphorothioate-modified oligonucleotides targeting the primary transcripts of the CD40, CD80 and CD86 co-stimulation molecules. The Control DC and the oligonucleotide-treated dendritic cells (iDC) are the study cell products in this proposal.

3.1.3 Leukapheresis Apparatus: This will be performed with the Fenwal CS3000 Plus cell collector, or equivalent, using a large bore double lumen catheter as peripheral venous access with total processing of approximately 10-12 liters per session. The device and its equivalents are FDA-approved for the procedures outlined herein to obtain purified leukocytes. Staff experienced with leukapheresis, contracted from the Central Blood Bank of Pittsburgh will perform these procedures.

3.1.4 Psychological Measures: The NEO-FFI is a 60 item paper and pencil questionnaire based on the five-factor theory of personality (Neuroticism, Extraversion, Openness, Agreeableness, and Conscientiousness). For this study we will examine the Neuroticism and Conscientiousness scales. The Beck Depression Inventory, 2nd edition (BDI-2) and the Beck Anxiety Inventory (BAI) are each 21 item paper and pencil questionnaires which have been widely used in psychiatric and medical populations.

3.2 Research Design and Methods 3.2.1 Setting/location of the study Systemic, physiologic and immunologic monitoring of patients prior to, during treatment cycle and post-treatment will take place in the CTRC clinic of Montefiore University Hospital of UPMC Health System (MUH-CTRC) under the supervision of the co-investigator physicians of this study and the nurses of the CTRC. Subjects will undergo leukapheresis in an outpatient setting at the MUH-CTRC or the University of Pittsburgh Cancer Center (UPCI) or the Central Blood Bank of Pittsburgh (depending on the most convenient location for each patient); receive the study dendritic cells in an outpatient setting at the MUH-CTRC; and undergo the remaining tests and procedures at the MUH-CTRC. Subjects will have approximately 16 visits at the locations described above, each visit lasting about 2-4 hours depending on what procedures are being performed at that particular visit. All results for each subject will be presented and discussed in an ongoing fashion at meetings held weekly at the UPCI outpatient clinic. Subjects will be monitored during the dendritic cell administration cycle; once every week following each dendritic cell administration for a period of nine weeks, then once a month for the remainder of the year (Refer to schematic cartoons in the Appendix, Section 6.8).

3.2.3 Autologous Control Dendritic Cell Vaccine Preparation Autologous DC will be generated from monocytes, derived from leukapheresis product. Leukapheresis will be performed at either of the following locations: 1) MUH-CTRC; 2) the UPCI Leukapheresis Unit; or 3) the downtown location of the Central Blood Bank of Pittsburgh. The product will be hand carried to the IMCPL located inside the Hillman Cancer Center in Shadyside by a nurse participating in the research study. At the time of procurement, immediately following leukapheresis, the sample will be coded by the nurse using the same code assigned to the patient during enrollment. At the IMCPL, monocytes will be separated by elutriation in a closed ELUTRA system. Monocytes will be cultured in the closed Aastrom Replicell System in the presence of IL-4 and GM-CSF to generate DC. On day 6 of culture, DC will be harvested and checked for viability and purity. An aliquot of freshly-generated DC will be used for the control DC vaccine preparation, while the remaining DC will be aliquoted into sterile cryovials and cryopreserved for preparation of subsequent vaccines. We have calculated that to prepare a vaccine containing 1 x 107 viable control dendritic cells or iDC (to be described below) for each delivery (One treatment defined as 1 x 107 dendritic cells injected at four intradermal sites anatomically-proximal to the pancreas) we will need a total of ~5 x 107 immature dendritic cells. This is the minimal cell number estimate, as additional aliquots of DC will be needed for testing prior to release of the vaccine for administration. The cells will be tested for viability, sterility (bacterial aerobic and anaerobic cultures and Gram stain), endotoxin level and mycoplasma as routinely performed by the IMCPL for cellular products used for human therapy at the UPCI. For each vaccine, the DC will be harvested, counted, adjusted into aliquots of 2.5 x 106 cells/mL in PBS with each aliquot and dispensed into a 1mL tuberculin syringe for future intradermal administration.

3.2.4 Oligonucleotide-treated (diabetes-suppressive) iDC Vaccine Preparation The same procedures as for the generation of control DC will be used to generate the iDC preparation with the inclusion of the antisense oligonucleotides at the same time as when GM-CSF and IL-4 will be added to the DC progenitors. The progenitors will be treated ex vivo with each of the antisense oligonucleotides to a final concentration of 3.3 μM according to SOP # CPL-0170 (Appended). On day 6 of culture, DC will be harvested and checked for viability and purity. After extensive washing to remove the remaining oligonucleotides from the culture medium, the iDC will be processed identically as above, dispensed into administration aliquots, and each aliquot will then be cryopreserved for future administrations.

3.2.5 Control and iDC Vaccine safety The vaccine will be prepared and administered to established type 1 diabetic patients meeting the criteria outlined in Section 4.0-4.1. The dendritic cell vaccines will be produced in the IMCPL, a cGMP facility which is in compliance with FDA recommendations for cellular products generated for patient therapy. At all times, the samples and the cell products will be identified by the same randomly-generated code assigned at the time of leukapheresis.

3.2.6. Safety evaluation: Initially, 15 patients (18-35 years of age) with established diabetes will be randomized to receive either the control dendritic cell vaccine (7/15 individuals) or the iDC (8/15 individuals) at the CHP GCRC. Randomization will be carried out using a macro (SUGI26) developed for the SAS statistics package. SUGI26 is a modification of a baseline adaptive randomization procedure and permits for unequal allocation ratios among multiple treatment groups for categorical covariates.

Following the establishment of the randomized patients into each treatment group, a patient may receive either of the two dendritic cell embodiments (control DC or iDC). These patients will receive 1 x 107 dendritic cells intradermally (four injections of 2.5 x 106 at four distinct sites anatomically-proximal to the pancreas) at the times illustrated in SECTION 3.2.1.1 and in the schematic cartoon (refer to the Appendix, Section 6.8) for a total of four vaccine administrations spaced every two weeks for a period of eight weeks. Per administration, we designate 4 unique intradermal injection sites inside the anterior abdominal wall perpendicularly-above the physical location of the stomach. These four sites will be within a quadrant of 3-4 square-inches. The cells will be delivered by a tuberculin syringe attached to a 27g-1/2 needle underneath a raised "bleb" of skin at each of the 4 individual injection sites. If there is no grade 3 or 4 toxicity observed following the first vaccine cycle in the DC recipients, successive vaccinations will be delivered as planned. Dose-limiting toxicities will be defined as equal to or greater than grade 2 with the following exceptions: chills, malaise and fever are not considered dose limiting. All grade 4 toxicities will be dose limiting, with the exception of lymphocytopenia. To protect patients against serious adverse effects of therapy the stopping rule will be observed, as described in Section 3.3.2 below. Following the leukapheresis procedure, the patient will be monitored for normoglycemia and if necessary, insulin will be administered as required to maintain normoglycemic levels. Glycemia will also be monitored at the end of each DC administration procedure and insulin can be administered to restore normoglycemia if necessary.

3.2.7 Dose-limiting toxicities:

The following are considered to be dose limiting toxicities (DLT's). If these toxicities are felt to be related to autologous dendritic cell vaccine administration, individual subjects will be immediately taken off study and no further injections will be given:

* ≥ Grade 2 or more bronchospasm,
* ≥ Grade 2 or more allergic reaction or generalized urticaria,
* ≥ Grade 2 or more autoimmune disease other than diabetes,
* ≥ Grade 2 injection site reaction due to vaccine or DTH testing,
* ≥ Grade 3 or 4 hematologic and non-hematologic toxicities
* Grade 2 toxicities that do not resolve within 5 days following the dendritic cell vaccine administration
* Dosing delays > 4 weeks

Therapy may be discontinued for the following reasons:

* Intercurrent illness that prevents further administration of autologous dendritic cell vaccine, including evidence of an infectious (bacterial/viral) disease
* Unacceptable adverse event(s),
* Patient decides to withdraw from the study, or
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator, nurse or attending physician(s).

3.3 DATA COLLECTION AND STATISTICAL CONSIDERATIONS 3.3.1 General Considerations This will be a safety trial to evaluate the safety and feasibility of administering a diabetes-suppressive dendritic cell vaccine based on autologous dendritic cells treated ex vivo with phosphorothioate-modified antisense oligonucleotides targeting the primary transcripts of the CD40, CD80 and CD86 co-stimulatory molecules. The vaccine will be given intradermally and each vaccine will contain 1 x 107 autologous dendritic cells. A total of 4 vaccines will be delivered to each eligible subject. A leukaphereses will be performed (14 days prior to the first vaccine) to ensure sufficient numbers of DCs.

The trial is designed to assure that the toxicity rate is acceptably low to warrant further study of the cell vaccine in efficacy trials.

4.5.1 CLINICAL TRIAL MONITORING

4.5.1.1 Reporting of Serious Adverse Events (SAE)

ADVERSE EVENTS: In general, all adverse events will be recorded and communicated to the safety officer, the PI and to the DSMB within 24 hours of occurrence. The safety officer will determine if the DSMB should meet under emergency session. Any non-serious adverse event reports will be submitted to the IRB within 24 hours of the DSMB meeting. The annual and final reports of the DSMB will also be submitted to the IRB and to the FDA within 48 hours of the meeting.

Reporting of Serious Adverse Events (SAE)

All (SAE) will be recorded on the standard toxicity sheets and reported to the FDA, the IRB, the DSMB safety officer, the Principal Investigator (Dr. Trucco) and/or Co-Investigators (Drs. Finegold, Whiteside or Giannoukakis) within 24 hours of occurrence. All treatment-emergent serious adverse events and pre-existing medical conditions which unexpectedly worsen during therapy will be recorded and reported as described immediately above (DSMB, DSMB safety officer, PI, FDA, IRB). All serious adverse events or deaths which occur beyond thirty (30) days and which are reasonably likely to be related to control or iDC administration will be reported within 24 hours of the event to the safety officer, the FDA and the full DSMB. Any serious or adverse events or deaths which occur within thirty (30) days of the last control DC or iDC administration will be reported identically. The safety officer will convene a full meeting of the DSMB within 24 hours of the occurrence of any SAE. The DSMB report will then be submitted to the IRB and the FDA no later than 48 hours following the occurrence of the SAE.

Serious is defined as described in 21 CFR 312.32 (a)

ELIGIBILITY:
Inclusion Criteria:

Patients with established type 1 diabetes mellitus who meet all inclusion criteria are eligible for enrollment in the study.

* All patients enrolled must be on insulin replacement therapy.
* Written informed consent conforming to the institutional guidelines obtained from the patient.
* Documented evidence of insulin-requiring type 1 diabetes of >5 years duration.
* Adequate immune competence, as indicated by positive reaction to one or more of the common DTH skin tests that are part of the Multitest CMITM test system (Pasteur-Merieux Connaught) and as indicated by the manufacturer. Also, proof of vaccination for tetanus (no more than 10 years must have elapsed between tetanus vaccination and the onset of this study).
* Age 18-35.
* Adequate hematologic function:

  * Absolute neutrophil count > 1,000/mm3
  * Absolute lymphocyte count > 1,000/mm3
* Hemoglobin > 9 gm/dl
* Platelets > 100,000/mm3
* Liver function tests:

  * Bilirubin (total) < 1.7 mg/dl
  * Alkaline phosphatase < 78 u/L (2 x ULN)
  * SGOT < 54 u/L (2 x ULN)
  * Lactic dehydrogenase < 180 u/L (2 x ULN)
* Kidney profile:

  * Serum electrolytes

    * Sodium 135-145 mEq/L
    * Potassium 3.5-5.0 mEq/L
    * Bicarbonate 21-28 mEq/L
    * Chloride 100-108 mmol/L
    * Serum creatinine <4.5 mg/dL (3 x ULN)
    * BUN 8-25 mg/dL
    * No prior history of radiation therapy, immunotherapy, or chemotherapy
    * Evidence of prior immunization to tetanus
    * Absence of HIV, HSV, HBV, HCV viral infections
    * At least four weeks since any prior radiation , immunotherapy or chemotherapy

Exclusion Criteria:

* One or more of the Eligibility Criteria are not met.
* A significant history or current evidence of cardiac disease including, but not limited to, congestive heart failure, coronary artery disease, angina pectoris, uncontrolled hypertension, serious arrhythmias; or myocardial infarction within the previous six months.
* Evidence of active infection requiring antibiotic therapy.
* History of other concurrent diseases.
* Pregnant or lactating women.
* Patients requiring systemic corticosteroids
* Any other immune disorder including but not limited to other autoimmune diseases like rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, or ankylosing spondylitis
* Pregnancy
* History of radiation therapy, immunotherapy, or chemotherapy
* Breastfeeding
* The following therapies cannot be administered while patients are undergoing treatment on this protocol:

  * radiation therapy
  * chemotherapy
  * corticosteroids (except when administered in life-threatening circumstances) other particle or cell vaccine therapies

At the time of screening, the patients will be tested for evidence of the following viral infections: HIV, HBV, HCV, herpes, CMV and EBV. In addition, female volunteers will be asked to provide documentation from their physician stating that they have not tested positive for the HPV viral infection. Only patients testing negative for ALL these viral infections will be further considered. Should any volunteer be excluded on grounds of positivity for any of these infectious agents, they will be immediately notified and strongly advised to consult their physician. The data and the records will be maintained under lock and in the study participation file of the volunteer until the volunteer confirms in writing that they have notified their physician. At that time, these specific data may be submitted to the patient's physician ONLY DIRECTLY BY THE VOLUNTEER upon written request to the study principal investigator or immediately destroyed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The trial is designed to assure that the toxicity rate is acceptably low to warrant further study of the cell vaccine in efficacy trials. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Trucco, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Harnaha J, Machen J, Wright M, Lakomy R, Styche A, Trucco M, Makaroun S, Giannoukakis N. Interleukin-7 is a survival factor for CD4+ CD25+ T-cells and is expressed by diabetes-suppressive dendritic cells. Diabetes. 2006 Jan;55(1):158-70. PMID 16380489
- [Result] Machen J, Harnaha J, Lakomy R, Styche A, Trucco M, Giannoukakis N. Antisense oligonucleotides down-regulating costimulation confer diabetes-preventive properties to nonobese diabetic mouse dendritic cells. J Immunol. 2004 Oct 1;173(7):4331-41. doi: 10.4049/jimmunol.173.7.4331. PMID 15383562
- [Derived] Phillips BE, Garciafigueroa Y, Engman C, Trucco M, Giannoukakis N. Tolerogenic Dendritic Cells and T-Regulatory Cells at the Clinical Trials Crossroad for the Treatment of Autoimmune Disease; Emphasis on Type 1 Diabetes Therapy. Front Immunol. 2019 Feb 6;10:148. doi: 10.3389/fimmu.2019.00148. eCollection 2019. PMID 30787930